CLINICAL TRIAL: NCT01848938
Title: Treatment of Stress Urinary Incontinence Via Smartphone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Eva Samuelsson, Associate professor, General Practitioner, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VisareNorr301811; JLL314561 (Other Grant/Funding Number: The County council of Jämtland); FAS2008-0952 (Other Grant/Funding Number: Swedish Council for Working Life and Social research); ALFVLL222081 (Other Grant/Funding Number: Västerbotten County Council (ALF))
Record Dates: First submitted 2013-04-26; First posted 2013-05-08 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Female Stress Urinary Incontinence
Keywords: female; stress urinary incontinence; treatment; pelvic floor muscle training; smartphone; internet; life style; eHealth
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone treatment (Active Comparator): Smartphone treatment with PFMT.
  Interventions: Behavioral: Smartphone treatment with PFMT
- Waiting list (No Intervention): Waiting list for three months. They receive the smartphone application after follow-up.

INTERVENTIONS:
Behavioral: Smartphone treatment with PFMT — A smartphone application with information on SUI, life style information, different programmes of PFMT with increasing severity, possibility to save statistics on training. The treatment period is three months
  Arms: Smartphone treatment

SUMMARY:
The purpose of this study is to determine whether treatment of stress urinary incontinence (SUI) via smartphone is effective.

DETAILED DESCRIPTION:
Female urinary incontinence (UI) is very common and affects up to one fourth of grownup women. It may reduce quality of life for those affected and costs for society are high. The most common type of urinary incontinence is SUI, i.e leakage when coughing, sneezing or jumping.

The recommended first line treatment is pelvic floor muscle training (PFMT)which leads to improvement or cure in two-thirds of patients. In addition, life style changes, such as weight loss when obese, smoking cessation and reduction of fluid intake if high is recommended.

There is a need for new , flexible and easily accessible treatment programmes for female urinary incontinence. In our previous study, we compared two treatment programmes for SUI without face-to-face contact: one internet based and one sent by post, both based on three months of PFMT. In this randomized controlled trial of 250 women aged 18-70 years, we found highly significant improvements (p<0.001) with large effect sizes (>0,8)concerning primary outcomes (symptoms and quality of life scores) but no significant differences between groups. Compared with the postal group, more participants in the internet group perceived they were much or very much improved (40.9% vs 26.5%, p<0.01, reported reduced usage of incontinence aids (59.5% vs 41.4%, p=0.02) and were satisfied with the treatment programme (84.8% vs 62.9%, p<0.001).

The selling of smartphones is increasing rapidly. About 75% of all cellphones sold in Sweden today are smartphones. Two million adults in Sweden have a smartphone. Many smartphone owners have at least one health app on their phone. Exercise, diet, and weight apps are the most popular types.

From our previous experience of an Internet-based programme, we have developed a treatment program designed for smartphone. The effect of the treatment programme will be evaluated after three months by comparing the effect in the "smartphone group" with the effect in the "waiting group".

Participants are consecutively recruited through our website. They answer an online screening survey with automated immediated response for initial screening of eligibility criteria. Informed consent and leakage diary (number of episodes of urinary leakage during 48 hours) are sent by post. After that, they answer a web questionnaire and finally they are interviewed by a researcher to confirm the diagnosis SUI and to ascertain that the patient is well informed of the study procedure.

Women are then randomized to either of the two groups. Women in the smartphone group get a smartphone application for iphone or android. Follow-up after three months with a web questionnaire and a leakage diary. After that the waiting group get their smartphone application.

We aim to recruit 120 women aged 18 and older via our website www.tät.nu. In the power calculation we assume that the improvement in the symptom score (ICIQ UI SF) and the QOL score (ICIQ luts QOL)in the smartphone group will be similar to the improvement we found in the postal group in our previous study. We also assume that the waiting group will improve in some extent.

To detect a difference between groups, power 80%, 2-side test and significance 0,05, group size as follow

ICIQ UI SF Smartphone group improves 2.9 (SD3,1) and waiting group 1,0 (SD2,0); 30 in each group

ICIQ luts QOL Smartphone group improves 4.6 (SD6,7) and waiting group 2.0(SD3.0), 35 in each group

PGI (patient´s global impression of improvement). 26,5% improves much or very much (smartphone) and 4% (waiting group):39 in each group

We expect a drop out rate of 33% and thus need approximately 120 persons, 60 in each group.

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence
* leakage once a week or more often
* duration of symptoms for at least 6 months
* motivation and time to perform a 12 week long treatment with pelvic floor muscle training
* ability to read and write Swedish
* asset to smartphone
* possibility to send and receive email and asset to printer
* accept to be randomized to one of two groups; a treatment group or a waiting list group

Exclusion Criteria:

* participation in our previous internet study
* pregnancy
* former incontinence surgery
* known malignancy in lower abdomen
* difficulties with passing urine
* visual blood in urine
* intermenstrual bleeding
* severe psychiatric diagnosis
* neurological disease with affection on sensibility in legs or lower abdomen
* urge incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Samuelsson, MD, PhD, Study Chair — Department of Public Health and Clinical Medicine, Umeå University
Locations (1):
- Umea University, Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asklund I, Samuelsson E, Hamberg K, Umefjord G, Sjostrom M. User Experience of an App-Based Treatment for Stress Urinary Incontinence: Qualitative Interview Study. J Med Internet Res. 2019 Mar 14;21(3):e11296. doi: 10.2196/11296. PMID 30869644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited community-dwelling women, from March 2013 to October 2014, through our website. Interested women filled out a questionnaire to determine whether they met the study criteria. Eligible women received a letter with informed consent and a 2-day leakage diary, and after returning this they also answered a web-based questionnaire.
Pre-assignment Details: Randomisation was performed by concealing the allocations in sequentially numbered, opaque, sealed envelopes. An independent administrator generated the allocation sequence and prepared 130 envelopes. The study coordinator opened one envelope for each participant and assigned an e-mail, with materials for the corresponding study group.
Groups:
- Smartphone Treatment: Smartphone treatment with PFMT.
  Smartphone treatment with PFMT: A smartphone application with information on SUI, life style information, different programmes of PFMT with increasing severity, possibility to save statistics on training. Possibility to set reminders. The treatment period is three months
Period: Overall Study
Arm/Group | Smartphone Treatment | Waiting List
Started | 62 | 61
Completed | 61 | 60
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Smartphone Treatment: Smartphone treatment with pelvic floor muscle training (PFMT).
  Smartphone treatment with PFMT: A smartphone application with information on SUI, life style information, different programmes of PFMT with increasing severity, possibility to save statistics on training. Possibility to set reminders. The treatment period is three months
- Total: Total of all reporting groups
Arm/Group | Smartphone Treatment | Waiting List | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (9.7) | 44.7 (9.1) | 44.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 62 | 61 | 123
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.0 (4.1) | 24.5 (4.4) | 24.2 (4.2)
Smoking [Number; unit: participants]
  smoker | 2 | 3 | 5
  non-smoker | 60 | 58 | 118
Education [Number; unit: participants]
  >=3 years at university level | 52 | 46 | 98
  <3 years at university level | 10 | 15 | 25
Parity [Number; unit: participants]
  nulliparous | 5 | 4 | 9
  not nulliparous | 57 | 57 | 114
Regular Medication [Number; unit: participants]
  on regular medication | 28 | 24 | 52
  no regular medication | 34 | 37 | 71
Usage of incontinence aids [Number; unit: participants] — Usage of incontinence aids during the last 4 weeks.
  participants
    No use | 6 | 10 | 16
    Less than once a week | 13 | 14 | 27
    1-3 times/week | 19 | 18 | 37
    >3 times/week, but not daily | 11 | 5 | 16
    1 aid a day | 9 | 10 | 19
    More than 1 aid a day | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: International Consultation on Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF)
Description: Three items on frequency, amount of leakage and overall impact. Scoring 0-21, higher values indicating increasing severity
Time Frame: baseline, three months
Population: intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 62 | 61
units on a scale
  baseline | 11.1 (3.0) | 11.0 (2.6)
  3 month follow-up | 7.0 (3.5) | 10.2 (3.2)
Statistical Analysis 1: Comparison: Smartphone Treatment vs Waiting List; analysis between groups; Test type: Superiority or Other; p < 0.001, Linear Mixed Models analysis

2. Primary Outcome: International Consultation on Incontinence Modular Questionnaire Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol)
Description: The instrument includes 19 items on the impact of the leakage. All items are scored 1-4 (not at all/never, slightly/sometimes, moderately/often, a lot/all the time). The overall score is 19-76, with higher values indicating increased impact on QOL.
Time Frame: baseline, three months
Population: intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 62 | 61
units on a scale
  baseline | 34.1 (6.1) | 34.8 (6.1)
  3 month follow-up | 28.8 (6.4) | 34.1 (6.7)
Statistical Analysis 1: Comparison: Smartphone Treatment vs Waiting List; analysis between groups; Test type: Superiority or Other; p = 0.005, Linear Mixed Models analysis

3. Secondary Outcome: Usage of Incontinence Aids
Description: Usage of incontinence aids during the last 4 weeks.
Time Frame: three months
Population: intention-to-treat analysis. Missing values at follow-up were replaced with the corresponding values at baseline (i.e., no change).
Measure: Number; unit: participants
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 62 | 61
participants
  No use | 23 | 14
  Less than once a week | 13 | 11
  1-3 times/week | 10 | 13
  >3 times/week, but not daily | 5 | 4
  1 aid a day | 8 | 12
  More than 1 aid a day | 2 | 6
Statistical Analysis 1: Comparison: Smartphone Treatment vs Waiting List; analysis between groups; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Patient Satisfaction
Description: A self-rated question about if the current treatment was sufficient, with three response options
Time Frame: three months
Population: Data for this outcome measure could only be collected for the smartphone treatment group.
Measure: Number; unit: participants
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 60 | 0
participants
  Yes, I am completely free of leakage | 5 |
  Yes, sufficient, although I am not completely free | 35 |
  No | 20 |

5. Secondary Outcome: Incontinence Episode Frequency (IEF)
Description: number of incontinence episodes per week
Time Frame: baseline, three months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: episodes per week
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 62 | 61
episodes per week
  baseline | 21.0 [10.5 to 28.0] | 17.5 [10.5 to 24.5]
  three month follow-up | 7 [0 to 14] | 14 [7 to 26]
Statistical Analysis 1: Comparison: Smartphone Treatment vs Waiting List; analysis between groups; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Patient's Global Impression of Improvement Scale (PGI-I)
Description: A self-rated question that asks about the change experienced after treatment with 7 response options, ranging from "very much better" to "very much worse".
Time Frame: three months
Population: intention-to-treat analysis. Missing values at follow-up were replaced with a neutral value (i.e., no change).
Measure: Number; unit: participants
Arm/Group | Smartphone Treatment | Waiting List
Number analyzed (Participants) | 62 | 61
participants
  very much better | 6 | 0
  much better | 28 | 3
  a little better | 22 | 9
  no change | 5 | 42
  a little worse | 0 | 6
  much worse | 0 | 0
  very much worse | 0 | 0
Statistical Analysis 1: Comparison: Smartphone Treatment vs Waiting List; analysis between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Smartphone Treatment | Waiting List
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 0/62 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No